



## **Consent Form for Participants**

## Full Title of Project: Remote monitoring use in suspected cases of COVID-19 (coronavirus): REMOTE-COVID trial

Name of Principal Investigator: Prof A Darzi

| | | | | Please initial box |
|---|---|---|---|---|
| 1. | I confirm that I have rea | | • | |
| | information sheet dated | | • | |
| | and have had the oppor | tunity to ask questions | s which have been | |
| | answered fully. | | | |
| | I understand that my pa | | | |
| | withdraw at any time, without giving any reason and without my | | | |
| | medical care or legal rights being affected. | | | |
| 3. | I understand that I will b | e wearing a wearable | monitoring patch. | |
| | I understand that I will b | • | | |
| | partake in an interview f | | | |
| | I understand that sections of any of my medical notes may be | | | |
| | looked at by responsible individuals from Imperial College London, | | | |
| | Chelsea & Westminster NHS Trust or from regulatory authorities | | | |
| | where it is relevant to my taking part in this research. | | | |
| | I give permission for these individuals to access my records that | | | |
| | are relevant to this research. | | | |
| 7. | 0, 0, 11, , | | | |
| | collected about me to be used to support other research in the | | | |
| | future, including those outside of the EEA. | | | |
| 8. | , , , , , , | | | |
| | remain anonymous; my name will not be used, nor any | | | |
| | information that could identify me. A transcription service may be | | | |
| | used to transcribe the information from the interview and all | | | |
| | interview data will be anonymised. | | | |
| 9. | I understand that what I say to the researcher will be recorded | | | |
| | using a digital voice recorder and saved on a computer at Imperial | | | |
| 10 | College London. | | | |
| 10 | . I understand what will h | appen and consent to | take part in the | |
| | above study. | | | |
| Name of Participant | | Signature | <br>Date | |
| Name of Person taking consent | | Signature | Date | |